CLINICAL TRIAL: NCT00626587
Title: Endobronchial Ultrasonography-Guided Transbronchial Needle Aspiration Increases the Diagnostic Yield of Peripheral Pulmonary Lesions : A Randomized Trial
Brief Title: EBUS-Guided TBNA Increases the Diagnostic Yield of Peripheral Pulmonary Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Meng-Chih Lin, Department of Internal Medicine, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CGMH-94-0101A; 96-0861B
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Last update posted 2008-02-29 (Estimated); Status verified 2005-01

CONDITIONS: Peripheral Pulmonary Lesions
Keywords: Endobronchial ultrasonography; Peripheral pulmonary lesions; Transbronchial needle aspiration; Probe location; Diagnostic yield; EBUS guided TBNA for peripheral pulmonary lesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Placebo Comparator): Conventional diagnostic procedures (transbronchial biopsy and bronchial washing) for peripheral pulmonary lesions
  Interventions: Device: Olympus NA-2C-1 Transbronchial needle aspiration (TBNA)

INTERVENTIONS:
Device: Olympus NA-2C-1 Transbronchial needle aspiration (TBNA) — The TBNA apparatus (Olympus NA-2C-1) is inserted through the working channel, and is advanced until it reaches the target lesion which is localized by EBUS. Negative manual suction is applied with the 20 ml syringe. The specimens are then smeared on glass slides and immersed in 95% alcohol. At least 3 aspirates per lesion are obtained.
  Other Names: TBNA apparatus (Olympus NA-2C-1) for bronchoscopic sampling

SUMMARY:
The diagnosis of peripheral pulmonary lesions(PPLs) remained a clinical challenge for physicians. Bronchoscope with sampling procedures was recognized as a useful method to obtain the correct diagnosis of PPLs. Conventional diagnostic procedures included transbronchial biopsy(TBB), bronchial washing(BW), or bronchial brushing, but the diagnostic yields were sometimes suboptimal. The diagnostic role of TBNA for PPLs remained to be determined, since many of the published studies were retrospective and had small sample size. This may explain the fact that TBNA was always underutilized for PPLs by bronchologists. With the popular application of EBUS-guided procedures in clinical setting, we performed EBUS-guided TBNA for PPLs. We want to determine whether EBUS-guided TBNA can improve the diagnostic rate of PPLs.

DETAILED DESCRIPTION:
The diagnostic yield of endobronchial ultrasonography (EBUS)-guided transbronchial needle aspiration (TBNA) for peripheral pulmonary lesions (PPLs) had not been evaluated. The diagnostic impact of TBNA when the EBUS probe was adjacent to lesions remained to be determined.

Here we designed a randomized, prospective study to evaluate : (1) The diagnostic yield of EBUS-guided TBNA in PPLs; (2) The role of TBNA when EBUS probe was adjacent to the lesions. Lesions not visible by bronchoscopy were defined as PPLs (no findings of endobronchial lesions, extrinsic compression, submucosal infiltration, or orifice narrowing). The TBNA apparatus (Olympus NA-2C-1) was inserted through the working channel, and was advanced until it reached the target lesion which was localized by EBUS. Negative manual suction was applied with the 20 ml syringe. The specimens were then smeared on glass slides and immersed in 95% alcohol. At least 3 aspirates per lesion were obtained. Using simple randomization with random digit table, we randomly assigned patients to undergo EBUS-guided TBB and BW or EBUS-guided TBNA, TBB and BW.

ELIGIBILITY:
Inclusion Criteria:

* Patients with peripheral pulmonary lesions (PPLs)

Exclusion Criteria:

* Repeated bronchoscopic examination
* Positive endobronchial lesions
* Negative EBUS findings

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2005-01; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The diagnostic yield of EBUS-guided TBNA in PPLs | Follow up of final diagnosis

SECONDARY OUTCOMES:
The role of TBNA when EBUS probe was adjacent to the lesions | Follow up of diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Lin Meng-Chih, MD, Principal Investigator — Chang Gung Memorial Hospital-Kaohsiung Medical Center
Locations (1):
- Chang Gung Memorial Hospital-Kaohsiung Medical Center, Niaosung Shiang, Kaohsiung, Taiwan

REFERENCES:
- [Derived] Chao TY, Chien MT, Lie CH, Chung YH, Wang JL, Lin MC. Endobronchial ultrasonography-guided transbronchial needle aspiration increases the diagnostic yield of peripheral pulmonary lesions: a randomized trial. Chest. 2009 Jul;136(1):229-236. doi: 10.1378/chest.08-0577. Epub 2008 Sep 23. PMID 18812446